CLINICAL TRIAL: NCT03440801
Title: A Randomized COmparison of LoNg-Term Vascular HealiNg bEtween Biodegradable -Polymer (BP) Versus Durable Polymer (DP) Everolimus Eluting Stents in Acute ST-Elevation Myocardial InfarCTion
Brief Title: A Randomized Comparison of Long-Term Healing Between Biodegradable- Versus Durable-Polymer Everolimus Eluting Stents in STEMI
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokorozawa Heart Center (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Masanori Taniwaki, MD, Tokorozawa Heart Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT1
Record Dates: First submitted 2018-02-12; First posted 2018-02-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Synergy (Experimental): Biodegradable-polymer everolimus-eluting stent Synergy
  Interventions: Device: Synergy; Device: Xience
- Xience (Active Comparator): Durable-polymer everolimus-eluting stent Xience
  Interventions: Device: Synergy; Device: Xience

INTERVENTIONS:
Device: Synergy — Biodegradable-polymer everolimus-eluting stent Synergy
Device: Xience — Durable-polymer everolimus-eluting stent Xience

SUMMARY:
This study aims to compare the acute thrombogenecity and frequency of neoatherosclerotic lesions and other aspects of long term arterial healing such as the frequency of malapposed and uncovered stent struts at 3 years among patients treated with either a biodegradable polymer everolimus-eluting stent (Synergy) or a durable polymer everolimus-eluting stent (Xience Alpine) for STEMI.

DETAILED DESCRIPTION:
DES use has significantly improved clinical outcomes as compared with bare metal stents (BMS), primarily through a notable reduction in the risk of repeat revascularisation. However, durable polymer DES have been associated with an increased risk of late and very late stent thrombosis and the anticipated development of in-stent neoatherosclerosis. In addition, in-vivo study suggest that different types of polymer among current DES might have different responses to acute thrombogenecity after stent implantation.

Patients with STEMI are associated with worse long-term clinical outcomes due to re-infarction and stent thrombosis throughout long-term follow-up. Underlying unstable lesion which includes ruptured plaque and thin-cap fibroatheroma behind stent strut is a predictor of neoatherosclerosis formation.

There is no dedicated randomized trial to comparing biodegradable-polymer versus durable polymer-DES in terms of acute thrombogenecity and long-term healing at 3 years after primary PCI.

Therefore this study is designed to compare the acute thrombogenecity and frequency of neoatherosclerotic lesions and other aspects of long term arterial healing at 3 years among patients treated with either a biodegradable polymer everolimus-eluting stent (Synergy) or a durable polymer everolimus-eluting stent (Xience Alpine) for STEMI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Primary PCI within 24 hours of symptom onset
3. ST-segment elevation of > 1mm in > 2 contiguous leads, or (presumably new) left bundle branch block, or true posterior MI with ST depression of >1mm in >2 contiguuoius anterior leads
4. Presence of at least one acute infarct artery target vessel with one or more coronary artery stenoses in a native coronary artery from 2.25 to 4.5 mm in diameter that can be covered with one or multiple stents

Exclusion Criteria:

1. Female ofchildbearing potential (age < 50 years and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy or hysterectomy.
2. Known intolerance to aspirin, clopidogrel, prasugrel, ticagrelor, heparin, stainless steel, cobalt chromium, platinum chromium, everolimus or contrast material
3. Inability to understand and provide informed consent
4. Currently participating in another trial before reaching first endpoint
5. Mechanical complications of acute myocardial infarction
6. Acute myocardial infarction secondary to stent thrombosis or restenosis
7. Planned surgery within 6 months of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period
8. Noncardiac comorbid conditions are present with life expectancy <3years or that may result in protocol noncompliance
9. History of bleeding diathesis or known coagulopathy
10. Use of oral anticoagulation
11. Age >90 years
12. LV-function at index procedure <=20%
13. Cancer under active treatment (chemotherapy)
14. Hemodynamic instability following primary PCI
15. Chronic kidey disease (Creatinine - Clearance < 30ml/min)
16. OCT technically not feasible (severe calcification, tortuosity)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Frequency of neoatheroslcerosis | 3 years
  Frequency of neoatherosclerosis lesion which is defined as the presence of a fibroatheroma or fibrocalcific plaques or macrophages within the neointima of a stented segment with a longitudinal extension of ≧ 1 mm at three years.

SECONDARY OUTCOMES:
Athero-thrombotic material area | initial day
  Athero-thrombotic material area (tissue protorusion + isolated intraluminal detect) within the stent strut after primary PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Tokorozawa Heart Center, Tokorozawa, Japan

REFERENCES:
- [Derived] Haner JD, Kakizaki R, Taniwaki M, Ohno Y, Yahagi K, Higuchi Y, Siontis GCM, Ando K, Stortecky S, Suzuki N, Watanabe N, Lanz J, Ueki Y, Otsuka T, Biccire FG, Sakurada M, Koskinas KC, Losdat S, Raber L. Low-Density Lipoprotein Cholesterol Levels and Neoatherosclerosis After STEMI: A Secondary Analysis of the CONNECT Randomized Clinical Trial. JAMA Cardiol. 2025 Dec 17:e254723. doi: 10.1001/jamacardio.2025.4723. Online ahead of print. PMID 41405905